CLINICAL TRIAL: NCT06447675
Title: Efficacy and Safety Evaluation of Hyperthermic Baths in the Treatment of Seizures in CDKL5 Deficiency Disorder: A Single-center, Self Control Trial
Brief Title: Efficacy and Safety Evaluation of Hyperthermic Baths in the Treatment of Seizures in CDKL5 Deficiency Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-111-002
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: CDKL5 Deficiency Disorder
Keywords: Hyperthermic Baths; Drug Resistant Epilepsy; CDKL5
MeSH Terms: conditions — CDKL5 deficiency disorder; Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperthermic Baths (Experimental): Patients with CDKL5 deficiency assigned to hyperthermic baths will have their body immersed in a hot water (40~42°C) bath for 20 min per session.
  Interventions: Other: Hyperthermic Baths

INTERVENTIONS:
Other: Hyperthermic Baths — The intervention will consist of 12 weeks of repeated (2x/day) 20-min body immersions.

SUMMARY:
The primary objective of this research is to study the efficacy and safety of hyperthermic baths as adjunctive therapy for reducing the frequency of seizures in CDKL5 deficiency.

DETAILED DESCRIPTION:
This project aims to include 8 participants, and evaluate the effectiveness and safety of hyperthermic baths in patients with CDKL5 deficiency through A single-center, preliminary feasibility clinical trial. It is expected to provide new therapeutic options for patients with CDKL5 deficiency with alternative treatment options.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CDKL5 deficiency, including molecular confirmation of a pathogenic or likely pathogenic CDKL5 variant and refractory seizures
* Male or female participants aged 6 months to less than 6 years
* Parent(s) or LAR willing to give written informed consent, after being properly informed of the nature and risks of the study and prior to engaging in any study-related procedures
* Failure to control seizures despite appropriate trial of 2 or more anti-seizure medications at therapeutic doses
* Have a history of at least 8 countable seizures per 4 weeks during the 8 weeks prior to screening. Countable seizures will be defined by the following:Seizures with or without impairment of consciousness with a clear motor component, including generalized tonic-clonic, focal to bilateral tonic-clonic, atonic, bilateral clonic, bilateral tonic, focal motor seizures with or without impaired awareness, or infantile spasms. Clusters of infantile spasms/tonic seizures will be counted as a single seizure.
* Participants should be on a stable regimen of anti-seizure medications for ≥ 4 weeks prior to the screening visit, without a foreseeable change in dosing for the duration of the DB phase.
* Vagus nerve stimulator (VNS) are permitted, but should be implanted for 1 year prior to screening and settings should be unchanged throughout the study.
* Parent/caregiver is able and willing to maintain an accurate and complete daily seizure eDiary for the duration of the study.

Exclusion Criteria:

* Any history of previous brain disease (trauma, etc.) that likely to precipitate seizures.
* Tissue damage (eczema, etc.) in the area where hyperthermic baths will be applied on the skin.
* Seizures associated with hyperthermic baths.
* Presence of any clinical condition that in the opinion of the principal investigator makes the patient not suitable to participate in the trial.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Seizure frequency (SF28) | Up to 3 month after hyperthermic baths
  Seizure frequency (SF28) is defined as seizure count per month (28-day) period. The SF28 is calculated as follows, where D=total number of days for which seizure information is collected for the specific 28-day interval:
  SF28=(Total number of seizures in D days/D)*28. In addition, the baseline seizure frequency is defined as SF28 in the baseline period. The seizure frequency in the treatment phase is defined as SF28 per month during the treatment period. Percent change in seizure frequency=100*(treatment SF28-baseline SF28)/baseline SF28.

SECONDARY OUTCOMES:
Seizure Responder Rate | Up to 3 month after hyperthermic baths
  The proportion of patients with a ≥ 50% reduction from Baseline in seizure frequency.
Seizure-free Days | Up to 3 month after hyperthermic baths
  Change in percentage of seizure-free days over the entire treatment phase as compared to the entire baseline phase. The number of seizure-free days was normalized to 84-day baseline and treatment phases for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No